CLINICAL TRIAL: NCT05243043
Title: Impact of an Interactive Maternal Resuscitation Navigation Application (MARINA) on Mothers' Experience During and After Premature Infant Resuscitation in the Delivery Room
Brief Title: Interactive Resuscitation Application for Mothers About to Experience Premature Infant Resuscitation
Status: Recruiting | Type: Observational
Sponsor: Stephanie Stewart (Other)
Responsible Party: Sponsor-Investigator, Stephanie Stewart, Associate Director, Nursing, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 202103564
Record Dates: First submitted 2022-01-13; First posted 2022-02-16 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Resuscitation
Keywords: Mothers' experience; Premature infant resuscitation; Post traumatic stress

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Mothers who experienced premature infant resuscitation in Labor and Delivery without the information provided by a computerized informational app.
- Intervention (future): Mothers who experienced premature infant resuscitation in Labor and Delivery with the information provided ahead of time by the computerized informational application.

SUMMARY:
The purpose of this study is to design, develop, validate and pilot test an interactive Maternal Resuscitation Navigation Application (MARINA) for the purpose of providing information and guidance about the expected events that a premature infant will experience during initial resuscitation upon delivery. This information will be shared via computer app prior to the time that the mother would be in distress due to active labor. The application will be pilot tested for functionality, usability and feasibility of future use and research in clinical settings. Focused aspects of the application will include simulated video of the active delivery environment, explanation of each team member's role in resuscitation and specific activities involved in premature infant resuscitation. To assure the application addresses key information mothers would desire, the application will include content developed with input from a consulting group of mothers who have experienced premature infant resuscitation in the delivery room. Additionally, prior research by the research team will inform the build of this application. The application will have the ability for mothers to choose whether to view close up procedures (bag/mask positive pressure oxygen delivery, intubation, line placement, etc.). She may alternatively select to only view the broader view of the room while listening to the description of activities occurring at that time. The mother will be able to choose her level of interactivity depending on her comfort level. The application will go through multiple levels of testing throughout the development process. After an iterative process, when the research team finds the application acceptable, a small group of consulting parents and experienced clinicians will review the application for functionality (ease of use) and content validity.

Aim 2: To pilot test the functionality, usability and feasibility of the interactive Maternal Resuscitation Navigation Application (MARINA) for future use and research in clinical settings to reduce maternal distress associated with premature infant resuscitation.

DETAILED DESCRIPTION:
AT THIS TIME, THE STUDY IS PROCEEDING WITH CONTROL GROUP ONLY. THE INTERVENTION PHASE OF THE STUDY WILL NOT BEGIN UNTIL A MODIFICATION WITH THE COMPLETED MARINA SOFTWARE APPLICATION IS SUBMITTED AND APPROVED BY THE BOARD. The purpose of this study is to design, develop, validate and pilot test an interactive Maternal Resuscitation Navigation Application (MARINA) for the purpose of providing information and guidance concerning premature infant resuscitation prior to the experience in the delivery room. The application will be pilot tested for functionality, usability and feasibility of future use and research in clinical settings.

Methods MARINA will be created by the University of Iowa Custom Solution and Integration (CSI) department, a division within the Information Technology Services. The application will use an interdisciplinary high-fidelity simulation video in a Labor & Delivery room setting as its core. Focused aspects of the video will include descriptions of the active delivery environment, explanation of each team member's role in resuscitation and specific activities involved in premature infant resuscitation. In order to establish content validity, the application will include content developed with input from a consulting group of mothers who have experienced premature infant resuscitation in the delivery room. Additionally, qualitative data and prior research by the research team will inform the build of this application.

The application will have the ability for mothers to choose whether to view close up procedures (bag/mask positive pressure oxygen delivery, intubation, line placement, etc.). She may alternatively select to only view the broader view of the room while listening to the description of activities occurring at that time. The mother will be able to choose her level of interactivity depending on her comfort level. The high-fidelity resuscitation will include voice over narration describing the steps and explaining key processes. By selecting a specific touch screen icon at crucial steps in the resuscitation process, the family can hear additional information from the narration or see additional angles of the procedure. The simulation will encourage the mother to be an active participant during her child's resuscitation with examples of the simulation mother asking question and receiving communication from the healthcare team caring for her infant. In order to evaluate usability and 'dose' of intervention, the application will include functionality to track which segments were accessed and amount of time spent by participant.

The application will go through multiple levels of testing throughout the development process. After an iterative process, when the research team finds the application acceptable, a small group of consulting parents and experienced clinicians will review the application for functionality (ease of use) and content validity.

Aim 2: To pilot test the functionality, usability and feasibility of the interactive Maternal Resuscitation Navigation Application (MARINA) for future use and research in clinical settings to reduce maternal distress associated with premature infant resuscitation.

Development and implementation of the application is targeted for mothers who are admitted to an inpatient OB unit for probable premature delivery.

Control group recruitment, enrollment and data collection In order to obtain baseline control group data to inform a future controlled trial, after informed consent, we will collect demographic data from the participant about their and their child, as well ask them to complete a survey. This will occur in 20 mother/infant dyad participants who were not exposed to MARINA prior to delivery, but experienced resuscitation of a premature infant. The control group survey will collect data for up to 40 subjects. The control group survey will include measures of traumatic stress including the Impact of Events Score - Revised (IES-R) and the Perinatal PTSD Questionnaire (PPQ-II). This will be a convenience sample of mothers whose newborn premature infants were delivered at UIHC between 24 and 32 weeks gestation. The newborn infants may or may not be currently admitted to the NICU at UI SFCH.

The research team will review the NICU census in Epic at least 4 days per week to identify infants who were born at UIHC between 24-32 weeks gestation. Emails will be sent to mothers of infants who meet inclusion/exclusion criteria with brief information about the study. If the mother chooses to participate in the study, she will be asked to click on a link that will take her to REDCap to review and sign the study consent form. After consent is completed, the study participant will be taken to the demographic data form to collect information about the participant and their child. Finally, upon completion of the demographic survey, participants will complete the research survey. The study information and link to participate will be sent again via email after 7 days of the initial email if the potential participant does not act on the invitation. Following the second email invitation, the potential participant will be contacted by phone by a research team member for the purposes of recruitment. The study team member will read the email invitation to the potential participant over the phone, then offer to re-send the recruitment email one last time if the participant chooses to participate.

Intervention group recruitment, enrollment and data collection L&D nursing and provider staff will be informed about the app and pilot study. Both nursing and provider staff will be presented with a brief PowerPoint presentation including information about the study including inclusion/exclusion criteria and how to reach a contact person for study recruitment. Additionally, there will be a sign placed near the L&D 'board' to remind staff about the study. On this sign, staff can write down the name of patients they have worked with who would meet inclusion/exclusion criteria. Study team members will check this list and review the antepartum and L&D census for potential participants each business day. Study personnel will be responsible for approaching potential participants. Intervention group will be a convenience sample of 20 women who are expected to deliver a premature infant between 24 and 32 weeks gestation. Data collected after delivery/post intervention will include 20 mother/infant group participants (20 mothers with up to 3 infants per mother (triplets, twins or singleton). The intervention group survey will collect data for up to 80 subjects.

Mothers of these infants who meet inclusion/exclusion criteria will be given a brief information sheet about the study after consultation with UIHC Neonatal Research nurses and the mother's care team. If the mother chooses to participate in the study, she will be asked to fill out the study consent form and answer demographic questions which will be recorded on a separate intake form (participant name, participant's birthdate, infant's name and birthdate, phone number and email address).

After enrolled in the study, the participant mother will be shown the MARINA. Study personnel will provide the mother with an iPad to use for viewing the application. Study personnel will instruct mother how to maneuver through the MARINA app. The mother will have access to the iPad for at least 30 minutes. Research personnel will go back to retrieve the device from the mother after 30 minutes or agreed upon time. If the mother has questions about what she viewed in the MARINA, the research team member or a member of her care team will answer these questions.

After the participant delivers her baby and experiences premature infant resuscitation in the delivery room, she will be scheduled to receive the post-delivery survey per email or text message 31 days or more post-delivery. Study personnel will track L&D and NICU census to determine when participant mothers deliver.

The survey for the intervention group will include questions about ease of use, the value of information provided in the application and one open text question for comments and suggestions, as well as the IES-R and PPQ-II measures.

Upon completion of the intervention group survey, participants will be invited to continue participation by participating in a brief interview regarding the usability of the application. One of the co-PIs will conduct the recorded, qualitative interviews. The interviews will be downloaded into secure password protected SharePoint site and transcribed word for word. After data validation, interview data will be coded by the co-PIs and at least one other research team member.

ELIGIBILITY:
Inclusion Criteria:

* Control group: English-speaking mothers, age 18 or older, delivered a premature infant at UIHC between 24- and 32-weeks and their infant born during this most recent gestation.

Exclusion Criteria:

* control group: Infant death, mothers who required general anesthesia at the time of delivery, active investigation by Department of Human Services, prisoners, twin gestation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Control group: 20 mother/infant dyads not exposed to MARINA prior to delivery, but experienced resuscitation of a premature infant. A convenience sample of mothers whose newborn premature infants were delivered at UIHC between 24 and 32 weeks gestation.
  Intervention group: A convenience sample of 20 women who are expected to deliver a premature infant between 24 and 32 weeks gestation, as well as their premature infant born post intervention.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Impact of Event Scale-Revised | Beginning 24 hours after a mother experiences her child's resuscitation until 65 days post the resuscitation.
  Impact of Event Scale - Revised (IES-R) is a tool that measures a participants risk for posttraumatic stress after experiencing an event. The IES-R consists of twenty two question items with a five point Likert scale ranging in response from zero to four, zero denotes low stress and four denotes high stress. The range of total scores is 0-88 with higher scores interpreted as a more stressful impact due to a traumatic event. A score of 24 has been determined to indicate a level of posttraumatic stress high enough for clinical concern.
Perinatal Post traumatic Stress Disorder Questionaire-II | Beginning 24 hours after a mother experiences her child's resuscitation until 65 days post the resuscitation.
  Perinatal Post traumatic Stress Disorder Questionaire-II (PPQ-II) is a 14-item tool measure assessing post-traumatic symptoms related to the childbirth experience, including intrusiveness or re-experiencing, avoidance behaviors and hyperarousal or numbing of responsiveness. The PPQ-II also contains one item pertaining to feelings of guilt. Response options include a five-point likert scale (scored 0 to 4). Mothers were instructed to provide responses that reflected their experience. The total possible score on the modified PPQ-II ranges from 0 to 56 with a higher score indicating a higher level of maternal distress.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Stewart, PhD, Principal Investigator — University of Iowa Stead Family Children's Hospital
Locations (1):
- University of Iowa Stead Family Children's Hospital, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Undecided